CLINICAL TRIAL: NCT05862675
Title: The Role and Mechanism of Immune Regulation in Acute Lung Injury in Children
Status: Withdrawn | Type: Observational
Why Stopped: Due to a time conflict in the research, the project research has been temporarily suspended.
Sponsor: Children's Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Bo liu, attending doctor, Children's Hospital of Chongqing Medical University
Other Study IDs: ChongqingMU
Record Dates: First submitted 2023-02-02; First posted 2023-05-17 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Acute Lung Injury
MeSH Terms: conditions — Acute Lung Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Collect blood, sputum or alveolar lavage fluid samples of subjects, extract RNA or DNA for relevant tests.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- experimental group: meeting the specific diagnostic criteria for acute Lung Injury
  Interventions: Diagnostic Test: RNA sequencing of blood samples
- control group: Healthy children

INTERVENTIONS:
Diagnostic Test: RNA sequencing of blood samples — Using omics techniques to detect blood samples from patients with acute lung injury and normal children, screen for marker genes related to immune cells in acute lung injury, and verify the protein expression of this molecule in tissues. Analyze the relationship between its phenotype and the degree of inflammation.
  Groups: experimental group

SUMMARY:
Acute lung injury is a highly prevalent disease in children, posing a serious threat to their health and causing economic burden on society and families. It has received high attention. Blocking the cascade immune inflammatory response that occurs in the respiratory tract and finding key targets for the prevention and treatment of acute lung injury has become an important challenge faced by the medical community. The pathogenesis of acute lung injury is complex, involving the combined action of multiple cells and cytokines in the immune system. Therefore, it is necessary to further study the function of immune cells and specific immune pathogenesis, providing new ideas and theoretical basis for clinical treatment of acute lung injury. The omics technology includes Genomics, Transcriptome, proteomics, metabolomics, etc. Through qualitative and quantitative analysis of changes in low molecular weight molecules or metabolites of biological samples, it provides a new way to find biomarkers and pathogenesis. We plan to study the peripheral blood of children with acute lung injury and healthy children, and use network analysis to screen for differential genes and related enrichment pathways in acute lung injury. We aim to explore the correlation between immune regulation and inflammatory repair in children with acute lung injury, and analyze the regulatory mechanisms between immune cells related to it. Provide assistance for clinical diagnosis and treatment.

DETAILED DESCRIPTION:
1. Inclusion criteria of the test group: (1) Meeting the specific diagnostic criteria for related lung diseases; (2) The factors of lung diseases were infection and sepsis;
2. Inclusion criteria of the control group: control 1: (1) Meeting the specific diagnostic criteria for related lung diseases; (2) The factors of lung diseases were non-infectious factors.

   Control 2: Healthy children
3. Exclusion criteria of the test group: (1) Patients with hemodynamic instability Patients with pulmonary hypertension;(2) Patients with congenital heart disease, congenital genetic metabolic disease, epilepsy, acute and chronic renal insufficiency, nephrotic syndrome, diabetes, et al.
4. The collection of clinical data includes: name, sex, age, hospitalization number, date of hospitalization, main diagnosis, course of disease, main examination and test results, medication, respiratory support, prognosis, etc.
5. Collect peripheral blood serum, sputum or alveolar lavage fluid samples for target sequencing.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of ALI/ARDS.
* Voluntary inclusion of researchers.

Exclusion Criteria:

* Patients with hemodynamic instability
* Patients with pulmonary hypertension
* Patients with congenital heart disease, congenital genetic metabolic disease, epilepsy, acute and chronic renal insufficiency, nephrotic syndrome, diabetes, etc.

Ages: 1 Year to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children aged 1-14 who were hospitalized in the Children's Hospital affiliated to Chongqing Medical University.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Degree of inflammation in acute lung injury through measure physiological parameter | an average of 1week
  The degree of inflammation includes changes in patient inflammatory indicators through measure physiological parameter.

SECONDARY OUTCOMES:
Expression of differential genes and proteins through gene sequencing | an average of 1week
  Detect patient gene expression through gene sequencing and analyze differential genes.

CONTACTS AND LOCATIONS:
Overall Officials: Zhou Mi, Master, Principal Investigator — Chongqing Medical University; Ding Fengxia, Doctor, Principal Investigator — Chongqing Medical University

IPD SHARING:
Plan to Share IPD: Undecided
If there is cooperation from other research centers in the future, this study will share patient clinical data and relevant clinical samples.

REFERENCES:
- [Background] Kumar V. Pulmonary Innate Immune Response Determines the Outcome of Inflammation During Pneumonia and Sepsis-Associated Acute Lung Injury. Front Immunol. 2020 Aug 4;11:1722. doi: 10.3389/fimmu.2020.01722. eCollection 2020. PMID 32849610
- See also: In order to have a more comprehensive understanding of this article, this link is used to view the original reference. — https://pubmed.ncbi.nlm.nih.gov/32849610/